CLINICAL TRIAL: NCT05425862
Title: Phase 1 Trial of Pidnarulex and Talazoparib in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Pidnarulex and Talazoparib in Patients With Metastatic Castration Resistant Prostate Cancer
Acronym: REPAIR
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrolment suspended to further assess supplementary non-clinical study data.
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20/019
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Castration Resistant Prostate Cancer (mCRPC)
MeSH Terms: interventions — CX 5461; talazoparib

STUDY DESIGN:
Intervention Model Description: This is phase I, open label, multicentre, dose-escalation study where both doses of talazoparib and pidnarulex will be escalated to define the MTD and RP2D for the combination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with both talazoparib and pidnarulex (Experimental): At the time of registration, patients will be assigned to the specific dose-schedule of talazoparib and pidnarulex depending on where the study is at in terms of dose-escalation or dose-expansion
  Interventions: Drug: Pidnarulex; Drug: Talazoparib

INTERVENTIONS:
Drug: Pidnarulex — Pidnarulex is a treatment that is designed to stop the action of a particular protein in the body called Polymerase I, that cancer cells rely on. Laboratory studies show that pidnarulex targets a process involving Polymerase I within cells, which can lead to a decrease in cancer growth. Pidnarulex has been shown to have some anticancer activity in ovarian cancer and haematological cancers.
  Other Names: CX-5461
Drug: Talazoparib — Talazoparib belongs to a class of drugs called PARP inhibitors, which is currently being used to treat various types of cancer. Talazoparib blocks the function of PARP, a protein that is involved in repairing DNA in cells. By stopping damaged DNA in cells from being repaired, this will lead to accumulation of DNA damage in the cancer cell and ultimately cancer cell death. Talazoparib has established anticancer activity in breast, ovarian and prostate cancers with underlying DNA repair defects. This class of drug have also been used in combination with other treatments such as radiation or chemotherapy to further increase cell death within the cancer.

SUMMARY:
This is phase I, open label, multicentre, dose-escalation study where both doses of talazoparib and pidnarulex will be escalated to define the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) for the combination. It is possible that either 1 or 2 RP2D of the combination will be defined at the end of the study. Patients with disease that is deemed to be amendable to repeated tumour biopsies will be invited to undergo optional paired biopsies: at baseline and Cycle 1 Day 9 + 3 days and at the time of progression. Pidnarulex will be given as an IV infusion on days 1 and 8 of a 28 day cycle and talazoparib will be taken once daily continuously. Disease status will be assessed at regular intervals by CT scans, radionuclide bone scans, and PSA. Throughout the study, safety and tolerability will be assessed and established procedures for management of toxicities will be applied

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥18 years of age and must have provided written informed consent.
2. Histologically confirmed adenocarcinoma of the prostate without neuroendocrine or small cell differentiation.
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
4. Patients must have had at least one prior treatment line of taxane (docetaxel) chemotherapy either in the hormone sensitive or castrate resistant setting unless the patient is deemed medically unsuitable for chemotherapy. If a patient has had docetaxel chemotherapy twice, this will be considered one line.
5. Patients must have progressed on a second-generation androgen receptor (AR) targeted agent (e.g. enzalutamide, abiraterone and/or apalutamide). Determination of disease progression on second-generation AR targeted agent will be made by the local Investigator.
6. Patients must have progressive disease (PD) for study entry. This is defined by Prostate Cancer Working Group 3 (PCWG3) as any one of the following:

   * PSA progression: minimum of two rising PSA values from a baseline measurement with an interval of ≥ 1 week between each measurement.
   * Soft tissue or visceral disease progression as per Response Evaluation Criteria in Solid Tumours (RECIST1.1) criteria
   * Bone progression: ≥ 2 new lesions on bone scan
7. The PSA value at screening should be ≥ 5ng/ml for all patients registered on the study.
8. At least 3 weeks since the completion of surgery or radiotherapy prior to commencing study treatment. Any clinically relevant sequelae from the surgery or radiotherapy must have improved to Grade 1 prior to Cycle 1 Day 1.
9. Prior surgical orchiectomy or chemical castration maintained on luteinizing hormone-releasing hormone (LHRH) analogue (agonist or antagonist). Patients without prior surgical castration must be currently taking and willing to continue LHRH analogue (agonist or antagonist) therapy throughout the duration of study treatment.
10. Serum testosterone levels ≤ 50ng/dL (≤ 1.75nmol/L) within 28 days prior to Cycle 1 Day 1.
11. Imaging evidence of metastatic disease documented with either bone scan or computerised tomography (CT) scan.
12. At least 3 weeks since completion of prostate cancer vaccine therapy, radiation therapy or systemic therapy prior to Cycle 1 Day 1.
13. Patients must have a life expectancy ≥ 24 weeks.
14. Male patients must use barrier contraception during treatment and for 3 months after the last dose of study drug when having sexual intercourse with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception.
15. Patients must be willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled assessments.
16. Patients must have adequate bone marrow, hepatic and renal function documented within 7 days prior to Cycle 1 Day 1, defined as:

    * Haemoglobin ≥100 g/L independent of transfusions (no red blood cell (RBC) transfusion in last 8 weeks)
    * Absolute neutrophil count (ANC) ≥1.2 x109/L
    * Platelets ≥120 x109/L
    * Total bilirubin ≤1.5 x upper limit of normal (ULN) except for patients with known Gilbert's syndrome where this applies to the conjugated bilirubin level.
    * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 x ULN if there is no evidence of liver metastasis or ≤5 x ULN in the presence of liver metastases.
    * Albumin ≥ 30 g/L
    * Adequate renal function: patients must have creatinine clearance (CrCl) estimated of ≥ 50 mL/min using the Cockcroft-Gault equation

Exclusion Criteria:

1. Extensive marrow disease defined by a "Super Scan" on bone scintigraphy or diffuse marrow infiltration on prostate specific membrane antigen (PSMA) positron emission tomography (PET).
2. Previous history or presence of brain metastases or leptomeningeal metastases. A scan to confirm the absence of brain metastases is not required if there is no clinical suspicion on history.
3. Surgery or radiotherapy within < 3 weeks prior to Cycle 1 Day 1 (except for palliative reasons). Patients must have recovered from effects of any major surgery.
4. Patients with symptomatic or impending cord compression unless adequately treated and clinically stable for ≥ 4 weeks.
5. Any prior exposure to platinums, poly (ADP-ribose) polymerase (PARP) inhibitors, mitoxantrone or cyclophosphamide.
6. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial lung disease on High Resolution CT scan or psychiatric illness/social situations that are likely to impede participation and/or compliance in the study.
7. Persistent toxicities (Common Terminology Criteria for Adverse Events [CTCAE] Grade 2) caused by previous cancer therapy, excluding alopecia.
8. Other malignancies within the previous 2-years that have a high risk of recurrence other than basal cell, squamous cell carcinomas of skin, melanoma in situ or other cancers that are unlikely to recur within 24 months.
9. Previous history of interstitial lung disease or non-infectious pneumonitis.
10. Patients with a history or clinical features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML).
11. Patients unable to swallow orally administered medications or with gastrointestinal disorders likely to interfere with the absorption of the study medication.
12. Resting Electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the Investigator (e.g., unstable angina, uncontrolled or symptomatic arrhythmia, congestive heart failure, corrected QT interval by Frederica [QTcF] prolongation >500ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
13. Known hypersensitivity to talazoparib or pidnarulex or any of the excipients of talazoparib or pidnarulex.
14. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV) 1/2. Serology only required if there is clinical suspicion on history. HIV-infected (HIV1/2 antibody-positive) patients may participate if they meet all the following eligibility requirements:

    * They must be on an anti-retroviral regimen with evidence of at least two undetectable viral loads within the past 6 months on the same regimen; the most recent undetectable viral load must be within the past 12 weeks They must have a CD4 count ≥250 cells/μL over the past 6 months on the same anti-retroviral regimen and must not have had a CD4 count <200 cells/μl over the past 2 years, unless it was deemed related to the cancer and/or chemotherapy-induced bone marrow suppression
    * For patients who have received chemotherapy in the past 6 months, a CD4 count <250 cells/μl during chemotherapy is permitted as long as viral loads were undetectable during this same treatment period
    * They must have an undetectable viral load and a CD4 count ≥250 cells/μL within 7 days prior to Cycle 1 Day 1
    * They must not be currently receiving prophylactic therapy for an opportunistic infection and must not have had an opportunistic infection within the past 6 months
15. Patients with active or uncontrolled infection, including hepatitis A, B or C. NOTE: Patients with controlled infection on antibiotic or antifungal therapy are eligible i.e. the patient should be afebrile for at least 72 hours and be haemodynamically stable.
16. Participation in another clinical study with an investigational product or another systemic therapy administered within 3 weeks prior to Cycle 1 Day 1.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-07-12 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The MTD is defined as the highest tolerable dose of pidnarulex when talazoparib is given at the highest tolerable dose and the highest dose of pidnarulex when talazoparib is given at the lowest dose (two MTDs will be estimated). | From study start to end of 2 years of recruitment period.

SECONDARY OUTCOMES:
Safety will be measured by serious adverse events (SAEs) and adverse events (AEs) assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0. | From the time of signing consent until 28 days after the last dose of protocol treatment.
Prostate Surface Antigen (PSA) response will be defined as a 50% or greater decrease in PSA from baseline to the lowest post-baseline PSA result. A second consecutive value obtained 4 or more weeks later confirms the PSA response. | From Cycle 1 Day 1 of treatment until the date of first documented progression, assessed up to 36 months.
Radiographic Progression Free Survival (rPFS) | From Cycle 1 Day 1 of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  The radiographic progression will be assessed by the Investigator per RECIST1.1 for soft tissue and PCWG3 for bone lesions. A patient who begins a new systemic anti-cancer treatment for clinical progression without documented radiographic progression will be censored at the time of initiation of new treatment. For patients alive who have no radiographic progression, the time will be censored at the date of last radiographic evaluation. The time will be censored at the date of treatment initiation for patients with no post-baseline radiographic evaluation.
Prostate Surface Antigen Progression Free Survival (PSA-PFS). | From Cycle 1 Day 1 of treatment until the date of first documented PSA progression or date of death from any cause, whichever came first, assessed up to 36 months.
Overall response (OR) is only applicable for the subset of patients with measurable disease by RECIST1.1. | From Cycle 1 Day 1 of treatment to the time of subsequent systemic anti-cancer treatment, assessed up to 36 months.
Overall survival (OS) | From Cycle 1 Day 1 of treatment to the date of death due to any cause, assessed up to 36 months.
Duration of Response Prostate Cancer Working Group 3 (DOR-PCWG3) | 12 weeks from Cycle 1 Day 1 of treatment to date of first documented radiographic progression. Assessed up to 36 months.
  (Patients who died of non-cancer causes without progression will be censored on the date of their last tumour assessment. A patient who begins a new systemic anticancer treatment for clinical progression without documented radiographic progression per RECIST1.1 for soft tissue and PCWG3 for bone lesions will be censored at the time of initiation of new treatment).
Treatment discontinuation at any time due to treatment related toxicity for each patient. | From study start to the end of study treatment. An average of 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Shahneen Sandhu, Principal Investigator — Peter MacCallum Cancer Research
Locations (5):
- Australia (5):
  - St Vincent's Hospital Sydney, Sydney, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Alfred Hospital, Prahran, Victoria

IPD SHARING:
Plan to Share IPD: No